CLINICAL TRIAL: NCT02806167
Title: A Study Into the Use of Post-Void Bladder Scanning as Part of a Clinical Algorithm for the Assessment of Patients With Suspected Acute Cauda Equina Syndrome
Brief Title: Post-void Bladder Scanning in Acute Cauda Equina Syndrome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Ethical approval declined
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RoyalDevon
Record Dates: First submitted 2016-06-15; First posted 2016-06-20 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2016-05

CONDITIONS: Polyradiculopathy
MeSH Terms: conditions — Polyradiculopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clinical algorithm (Experimental): This is a single arm study. All eligible patients will be subject to our clinical algorithm.
  Interventions: Other: Clinical algorithm

INTERVENTIONS:
Other: Clinical algorithm — Patients presenting with suspected acute CES will be assessed in accordance with the algorithm previously outlined.

SUMMARY:
Expedient diagnosis and management of acute cauda equina syndrome (CES) is essential to prevent long-term neurological sequelae for these patients. The clinical diagnosis of CES is confirmed using magnetic resonance imaging (MRI). However the clinical features of CES (secondary to bladder and bowel sphincter dysfunction) are variable and are common presenting features of other pathologies of the bladder and bowel, therefore most patients who undergo MRI for suspected CES have no compressive lesion evident on the MRI, excluding the diagnosis of CES. Urgent MRI scanning performed out of hours is therefore often unnecessary, however, the morbidity to the patient due to a delay in diagnosis is so significant that urgent MRI scanning is the current gold standard and duty of care in all cases of suspected CES. More objective methods of assessing patients with suspected acute CES could allow rationing of out of hours MRI scanning and reduce inappropriate admission without impacting patient safety.

The aim of this study is to evaluate the effectiveness of a clinical algorithm which utilises digital rectal examination and ultrasound bladder scanning to stratify patients into high and low risk groups. Patients considered high risk will be admitted and sent for urgent MRI, whereas low risk patients will be discharged and undergo MRI scan within 5 days of presentation.

DETAILED DESCRIPTION:
All patients with suspected CES will be seen and assessed by a member of the on-call team i.e. either a spinal fellow, spinal SpR, orthopaedic SpR or junior doctor, on presentation. Clinical features will be documented and stored in the patient notes. This document will then be photocopied for use in the study. Digital rectal examination will be performed to assess anal sphincter tone, voluntary control (anal contraction) and sensation of sharp and light touch with a chaperone present. Those with abnormal perianal sensation will be admitted and referred for urgent MRI. (NB: For the purposes of this study, these patients will also undergo pre and post-micturition bladder scans in order to allow the correlation between perianal sensation and residual urine volume to be assessed thoroughly.)

Bladder scanning will be used to measure pre and post-micturition residual urine volume in patients with normal perianal sensation. The on-call spinal registrar, fellow or consultant will conduct the bladder scanning using the BARDSCAN IIs ultrasound device. Patients with residual urine volume greater than 100ml will be admitted and referred for urgent MRI. Patients with normal perianal sensation and residual urine volume less than 100ml however will be discharged and receive an MRI scan as an outpatient within 5 days of presentation. These patients will be advised that if there is any progression of their symptoms that they should re-attend hospital. Any patient who re-attends, whilst waiting for their out-patient MRI, will be admitted for an urgent MRI.

Assessment of patients unable to void following pre-micturition bladder scan will depend upon bladder volume. Those measuring greater than 100ml will be catheterised and sent for MRI, whereas patients with less than 100ml will be encouraged to try again in 1 hour. Patients who fail to void at this time will also be catheterised and sent for MRI.

Patient Follow-up All patients will be followed-up by the consultant responsible for their care. Patients operated on for confirmed CES will be seen in clinic at six weeks and six months following surgery (or as required). Patients who do not require surgery will be seen in the next available clinic (usually within two weeks). Any unfortunate patients who continue to experience bladder and/or bowel dysfunction as a complication of CES will be referred to urology, urogynaecology, neurology and/ or colorectal services as appropriate.

Data Synthesis, Management and Analysis A pro forma will be used to assess all cases of suspected CES. This will be completed as part of the initial assessment by a member of the on-call spinal team and stored in the patient's notes. Demographic data will also be collected. These documents will be photocopied from the notes and data transferred to an Excel spread sheet and stored on an RD&E NHS password protected computer. Hospital number will serve as the only patient identifier. Photocopies will be stored in the spinal research office, which will be locked when not in use. Data will be stored for ten years following the end of the study period before destruction.

Statistical analysis will be carried out using IBM SPSS Statistics v21 for Mac. Descriptive statistics will be calculated and comparisons of means carried out according to the distribution of data. The sensitivity and specificity of our proposed diagnosis algorithm, as well as positive predictive values, will be calculated according to a 2x2 table. For between groups analyses ANOVA will be used and for testing differences between patients with and without post-residual volume >100ml, an independent t-test will be performed. A p value below 0.05 was considered to be statistically significant.

Dissemination of Results To the best of our knowledge this is the first study to investigate the use of post-micturition bladder scanning as part of a clinical algorithm for patients with suspected acute CES. It is the intention of the investigators to disseminate the outcomes of this study to regional, national and international scientific peer groups.

Authorship, accountability and acknowledgement will follow guidance as outlined by International Committee of Medical Editors. For core protocol publications (reporting on primary and secondary objectives of the trial), the protocol team serves as the writing team, usually with the protocol chair as lead author. For cross-protocol publications, with the permission of lead investigator, other team members may act as writing team and may include other additional authors as appropriate. Additional authors may include other investigators, usually members of trial staffs or inter-departmental collaborators, and/or site investigators. The principal investigator or other protocol team members may present data at scientific meetings.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected CES
* Minimum age 18 years.
* Both sexes
* Able to provide informed consent for their data to be included in the study

Exclusion Criteria:

* Patients with pre-existing urinary tract pathologies (neuropathic bladder, urologic pathologies or surgery, history of urinary incontinence.)
* Under age of 18 years.
* Patients with urinary catheter for whatever reason.
* Prisoners.
* Patients unable to provide informed consent for themselves.
* Previous spinal surgery
* Patients with urinary tract infections
* Patients with pre-existing neurological conditions affecting:
* Central nervous system such as multiple sclerosis
* Peripheral nervous system such as diabetic neuropathy, B12 deficiencies, thyroid abnormalities
* Autonomic nervous system such as multiple system atrophy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2019-09 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Successful risk stratification | 36 months
  The study will aim to stratify patients into high and low risk of CES though implementation of an algorithm which uses bladder scanning. The algorithm will be deemed successful if no patients are missed.

SECONDARY OUTCOMES:
Correlation between clinical assessment and residual urine volume | 36 months
  We will measure pre and post-micturition bladder urine volumes in all consenting patients with normal and abnormal perianal sensation in order to allow the correlation between clinical assessment and residual urine volume to be assessed thoroughly.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Stokes, FRCS, Principal Investigator — Royal Devon and Exeter NHS Foundation Trust
Locations (1):
- Royal Devon and Exeter NHS Foundation Trust, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No